CLINICAL TRIAL: NCT00732771
Title: A Pilot, Single-blind, Forced-titration Study to Assess the Hemodynamic and Hormonal Effects, Safety and Tolerability of the Aldosterone Synthase Inhibitor LCI699 in Patients With Primary Hyperaldosteronism
Brief Title: Proof-of-concept for the Aldosterone Synthase Inhibitor LCI699 in Patients With Primary Hyperaldosteronism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CLCI699A2206
Record Dates: First submitted 2008-08-05; First posted 2008-08-12 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Primary Hyperaldosteronism
Keywords: primary hyperaldosteronism; hypokalemia; hypertension; aldosterone synthase inhibitor
MeSH Terms: conditions — Hyperaldosteronism; Hypokalemia; Hypertension | interventions — Osilodrostat

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- LCI696 1mg bid (Experimental)
  Interventions: Drug: LCI699

INTERVENTIONS:
Drug: LCI699

SUMMARY:
The purpose of this study is to determine if LCI699, thorough reductions in aldosterone, can lower BP in patients with Primary hyperaldosteronism.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary hyperaldosteronism (PH) within the last 3 years, either with or without an aldosterone producing adenoma (APA).
* Hypertension at screening

Exclusion Criteria:

* Persistent hypokalemia
* Renal impairment
* Significant hepatic disease
* Any surgical or medical condition which may significantly alter the absorption, distribution, metabolism or excretion of any drug substance

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure over a 7-week forced titration treatment period | 7 weeks

SECONDARY OUTCOMES:
Plasma and urine hormone levels and electrolytes, diastolic blood pressure and drug pharmacokinetics over a 7-week forced titration treatment period | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigator site
Locations (1):
- Novartis Investigator Site, France, France

REFERENCES:
- [Derived] Schumacher CD, Steele RE, Brunner HR. Aldosterone synthase inhibition for the treatment of hypertension and the derived mechanistic requirements for a new therapeutic strategy. J Hypertens. 2013 Oct;31(10):2085-93. doi: 10.1097/HJH.0b013e328363570c. PMID 24107737
- [Derived] Amar L, Azizi M, Menard J, Peyrard S, Watson C, Plouin PF. Aldosterone synthase inhibition with LCI699: a proof-of-concept study in patients with primary aldosteronism. Hypertension. 2010 Nov;56(5):831-8. doi: 10.1161/HYPERTENSIONAHA.110.157271. Epub 2010 Sep 13. PMID 20837883